CLINICAL TRIAL: NCT04486040
Title: Closed Suction Drainage After Revision Hip Arthroplasty - Prospective Randomized Study
Brief Title: Closed Suction Drainage After Revision Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof A Gruca Teaching Hospital (Other)
Responsible Party: Principal Investigator, Bartosz Paweł, M.D., Ph.D. Principal Investigator, Prof A Gruca Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GrucaTH
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Hip Osteoarthritis; Bleeding
Keywords: Hip; Revision; Arthroplasty; Drainage
MeSH Terms: conditions — Osteoarthritis, Hip; Hemorrhage | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drainage group (Active Comparator): Patients with drainage after hip revision arthroplasty
  Interventions: Procedure: Drainage
- No-drainage group (Active Comparator): Patients without drainage after hip revision arthroplasty
  Interventions: Procedure: No-drainage

INTERVENTIONS:
Procedure: Drainage — Use of the suction drainage after hip revision arthroplasty
  Arms: Drainage group
Procedure: No-drainage — Patients without drainage after surgery
  Arms: No-drainage group

SUMMARY:
Prospective, randomized trial. 40 patients who underwent revision hip arthroplasty, divided in to two groups with or without drainage. All patients was assessed with ultrasonography on 3rd day after surgery. Bleeding, need for blood transfusion and laboratory test was analyzed after surgery. Patients was assessed with Harris Hips Score and Visual Analog Scale after surgery.

DETAILED DESCRIPTION:
Inclusion criteria: aseptic loosening, head or insert damage, girdlestone hip. Exclusion criteria: septic loosening, primary or secondary coagulopathy, renal or hepatic failure, thromboembolism in past history. At the end of operation information of drainage was get out from the envelope. On 3rd day all patient get ultrasonography with level of fluid in the joint and hematoma in soft tissue measurement. We analyzed hemoglobin, C-reactive protein, erythrocyte sedimentation rate on 1st and 3rd day after surgery. Visual analog scale was taken on 3rd day after surgery and Harris Hip Score 6 weeks after.

ELIGIBILITY:
Inclusion Criteria:

* aseptic loosening,
* head or insert damage,
* girdlestone hip

Exclusion Criteria:

* septic loosening,
* primary or secondary coagulopathy,
* renal or hepatic failure,
* thromboembolism in past history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Hematoma size | 3 days after surgery
  Level of fluid at endoprosthesis neck in ultrasonography
Hemoglobin level | 3 days after surgery
  Hemoglobin level after surgery on 1st and 3rd day after surgery
Blood loss | 1 day after surgery
  Assessing blood loss with use of Gross formula
Reinfection | 2 years after surgery
  Number of patients with infection after surgery performed in the study

SECONDARY OUTCOMES:
Soft tissue hematoma | 3 days after surgery
  Note hematoma formation in soft tissue after surgery (ultrasonography)
C-reactive protein level | 3 days after surgery
  Level of C-reactive protein after surgery
Blood transfusion | 5-14 days after surgery
  Number of patients who need blood transfusion after surgery
Visual Analog Scale | 3 days after surgery
  Level of pain after surgery, 1- no pain; 10- "the worst pain you ever had"
Harris Hip Score | 6 weeks after surgery
  Clinical outcome after surgery, 0-100 points; 100 points the best score

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Bartosz, Principal Investigator — Gruca Teaching Hospital, Centre of Postgraduate Medical Education in Otwock

IPD SHARING:
Plan to Share IPD: No